CLINICAL TRIAL: NCT01454986
Title: A Phase 1, Randomized, Blinded, Placebo-Controlled, Single-Administration, Sequential-Cohort Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of ALXN1007 in Healthy Subjects
Brief Title: Study to Evaluate Safety, Tolerability, PK and PD of ALXN1007 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C11-002
Record Dates: First submitted 2011-10-07; First posted 2011-10-19 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Healthy
Keywords: Healthy subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Cohort 1 (Active Comparator): 0.06 mg/kg ALXN1007
  Interventions: Drug: ALXN1007; Other: Placebo
- Cohort 2 (Active Comparator): 0.1 mg/kg ALXN1007
  Interventions: Drug: ALXN1007; Other: Placebo
- Cohort 3 (Active Comparator): 0.3 mg/kg ALXN1007
  Interventions: Drug: ALXN1007; Other: Placebo
- Cohort 4 (Active Comparator): 1.0 mg/kg ALXN1007
  Interventions: Drug: ALXN1007; Other: Placebo
- Cohort 5 (Active Comparator): 3.0 mg/kg ALXN1007
  Interventions: Drug: ALXN1007; Other: Placebo
- Cohort 6 (Active Comparator): 6.0 mg/kg ALXN1007
  Interventions: Drug: ALXN1007; Other: Placebo
- Cohort 7 (Active Comparator): 10.0 mg/kg ALXN1007
  Interventions: Drug: ALXN1007; Other: Placebo

INTERVENTIONS:
Drug: ALXN1007 — Single dose, IV
Other: Placebo — Single dose, IV

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, PK and PD of a single-dose of ALXN1007 in healthy volunteers.

DETAILED DESCRIPTION:
All subjects will be screened for eligibility after providing signed informed consent. Once a subject is determined to be eligible, the subject will be vaccinated with the quadrivalent meningococcal conjugate vaccine at least two weeks prior to dosing, if applicable. A total of 7 dose cohorts will be enrolled sequentially and randomized to receive ALXN1007 or placebo. Subjects will receive ALXN1007 or placebo at the clinic and be kept at the clinic for a total of 4 days for observation and completion of the required study tests.

The subjects will return for 8 additional clinic visits to complete the required study tests over the next 86 days. The total duration of the study is 90 days from the day of dosing with ALXN1007 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals 25 to 55 years of age with documented vaccination with MCV4.

Exclusion Criteria:

* Abnormal renal or liver function.
* History of meningococcal disease.
* History of Guillain-Barre syndrome.
* Known infection with HIV or Hepatitis B or C.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a single dose of ALXN1007. | Up to 90 days
  Safety and tolerability of a single dose of ALXN1007 assessed by physical exam, vital signs, ECG, immunogenicity, lab analysis and adverse events.

SECONDARY OUTCOMES:
PK parameters of ALXN1007 | Up to 90 days
  Estimate PK parameters of ALXN1007 using standard measures for these parameters.
PD parameters of ALXN1007 | Up to 90 days
  Identify PD effects of ALXN1007 by assessing standard complement measures for these parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- PAREXEL Baltimore EPCU, Baltimore, Maryland, United States